CLINICAL TRIAL: NCT07248839
Title: A Phase 1, Multi-center, Open-label, Single-dose Study to Assess the Pharmacokinetics and Safety of BMS-986435 in Participants With Normal Hepatic Function and Participants With Mild and Moderate Hepatic Impairment
Brief Title: A Study to Assess the Drug Levels and Safety of BMS-986435 in Participants With Normal Hepatic Function and Participants With Different Degrees of Hepatic Impairment
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CV029-1017
Record Dates: First submitted 2025-11-18; First posted 2025-11-25 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Healthy Volunteers; Hepatic Impairment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Arm A (Experimental): Mild Hepatic Impairment
  Interventions: Drug: BMS-986435
- Arm B (Experimental): Moderate Hepatic Impairment
  Interventions: Drug: BMS-986435
- Arm C (Experimental): Matched participants with normal hepatic function
  Interventions: Drug: BMS-986435

INTERVENTIONS:
Drug: BMS-986435 — Specified dose on specified days
  Other Names: MYK-224

SUMMARY:
The purpose of this study is to determine the pharmacokinetic and safety of BMS-986435 in participants with normal hepatic function and participants with different degrees of hepatic impairment

ELIGIBILITY:
Inclusion Criteria:

* Participant must have documented LVEF ≥ 60% (2D biplane Simpson's Method) and absence of cardiac abnormality.
* Participant must have body weight of > 50 kg and BMI of 18.0 kg/m2 through 40 kg/m2, inclusive, at screening.
* Participants must have adequate renal function at screening as evidenced by an eGFR > 60 mL/min/1.73 m2 for participants calculated with the CKD-EPI Creatinine Equation (2021).

Exclusion Criteria:

* Participants must not have history of or current uncontrolled or unstable clinically significant disorder, condition, or disease that, in the opinion of the investigator and CRO MM, would pose a risk to participant safety or interfere with the study evaluation, procedures, or completion.
* Participants must not have head injury in the last 2 years, intracranial tumor, or aneurysm.
* Participants must not have history of malignancy of any type, except in situ cervical cancer >5 years prior to the screening visit or surgically excised non-melanomatous skin cancer >2 years prior to the screening visit.
* Participants must not have History of heart disease (including coronary artery disease, heart failure/LV systolic dysfunction, cardiomyopathy, or clinically significant structural disease).
* Other protocol defined inclusion/exclusion criteria applies.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-12-15 (Estimated); Primary Completion 2026-04-06 (Estimated); Study Completion 2026-04-06 (Estimated)

PRIMARY OUTCOMES:
Maximum observed concentration (Cmax) | Up to Day 45
Area under the concentration-time curve from time zero to time of last quantifiable concentration AUC(0-T) | Up to Day 45
Area under the concentration-time curve from time zero extrapolated to infinite time AUC(INF) | Up to Day 45

SECONDARY OUTCOMES:
Number of participants with adverse events (AEs) | Up to Day 45
Number of participants with serious adverse events (SAEs) | Up to Day 45
Time of maximum observed concentration (Tmax) | Up to Day 45
Half-life (T-HALF) | Up to Day 45
Apparent total body clearance (CLT/F) | Up to Day 45
Apparent volume of distribution at terminal phase (Vz/F) | Up to Day 45

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb

IPD SHARING:
Plan to Share IPD: Yes
BMS will provide access to individual anonymized participant data upon request from qualified researchers, and subject to certain criteria.
  Additional information regarding Bristol Myers Squibb's data sharing policy and process can be found at: https://www.bms.com/researchers-and-partners/clinical-trials-and-research/disclosure-commitment.html
Supporting Information: Study Protocol, SAP, CSR
Time Frame: See Plan Description
Access Criteria: See Plan Description
URL: https://www.bms.com/researchers-and-partners/clinical-trials-and-research/disclosure-commitment.html

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.BMSClinicalTrials.com